CLINICAL TRIAL: NCT02948738
Title: Asthma Inpatient Research on Education: A Randomized Clinical Trial
Brief Title: Asthma Inpatient Research on Education
Acronym: AIREd
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Waheeda Samady, MD, Physician, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ChildrensMemorialH
Record Dates: First submitted 2016-10-27; First posted 2016-10-28 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Asthmatic Attack

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interactive Education (Experimental): Interactive asthma education
  Interventions: Behavioral: Interactive Asthma Education
- Standard Education (Active Comparator): Standard asthma education
  Interventions: Behavioral: Standard Asthma Education

INTERVENTIONS:
Behavioral: Interactive Asthma Education — Active participation to develop asthma action plan and teach back cycles for asthma inhaler teaching/training
  Arms: Interactive Education
Behavioral: Standard Asthma Education — Basic review of asthma action plan and inhaler use
  Arms: Standard Education

SUMMARY:
Children with asthma are admitted for asthma attacks very frequently in the U.S. The families and children are given basic education about asthma but studies are needed to improve this education so that it makes a meaningful difference in health outcomes and asthma care. This study compares two inpatient education models for children hospitalized with asthma.

DETAILED DESCRIPTION:
The current standard is to review an asthma action plan with families and to review inhaler medication administration. In this study, investigators will be assigning families to either a control (current standard education) or and intervention group. In the intervention group, participants will receive interactive education based on learning theories that are thought to enhance long term memory. Participants in the interactive group will build their own action plan using colored templates and pictures. Participants will also learn to use their inhaler using teach-back methodologies. Investigators will then compare the two groups in terms of ER visits, hospitalizations, family confidence in managing asthma, asthma knowledge, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma

Exclusion Criteria:

* Active Cardiac Disease
* Speaks language other than English or Spanish

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
ER visits | 1 year
  Number of ER visits in the year after education

CONTACTS AND LOCATIONS:
Overall Officials: Waheeda Samady, MD, Principal Investigator — Northwestern University and Lurie Children's Hospital
Locations (1):
- Ann and Robert H. Lurie Childrens Hosptial of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No